CLINICAL TRIAL: NCT06859021
Title: Validation of the HAR Score for Prioritization of Patients Calling the Emergency Medical Service for Chest Pain by Emergency Call Dispatcher : Reg-HAR Study
Brief Title: Validation of the HAR Score for Prioritization of Patients Calling the Emergency Medical Service for Chest Pain by Emergency Call Dispatcher
Acronym: Reg-HAR
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2024-S01-08
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chest Pain
Keywords: Chestpain; HAR score; Emergency call
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- call for chest pain: patients who call for chest pain
  Interventions: Other: follow up call

INTERVENTIONS:
Other: follow up call — A follow-up call is made to the patient 30 days (+ 5 days) after inclusion to check for the occurrence of an Major Cardio Vascular Event.

SUMMARY:
The lifetime prevalence of chest pain in the general population is 20-40%. The etiologies to be evoked from the outset of management are those of cardiovascular origin, such as acute coronary syndrome (ACS) and pulmonary embolism. ACS is responsible for almost 20% of deaths. Delay in treatment is a major prognostic factor, given the importance of coronary reperfusion.

In France, one of the first contacts with the healthcare system is the medical regulation assistant (MRA) at the Centre 15. His or her role is to prioritize the call according to the identification of immediate signs of seriousness, and if necessary, to decide autonomously to send a rescue team before medical regulation. Depending on the reason for the call and any signs of seriousness, it prioritizes the call according to the expected response time. In line with current recommendations, all calls for chest pain should be answered by an emergency medical dispatcher (EMR) within 5 minutes. However, 60-90% of chest pain calls are not of cardiovascular origin. Their prioritization could therefore be re-qualified for longer response times.

Given the frequency of this type of call, a more efficient MRA referral strategy is needed. To achieve this, decision-support tools would be essential.

The performance of the HAR (History, Age and Risk Factors) score has been recently explored, derived from the HEART score, in a previous single-center prospective study in 2019. It stratifies the risk of a major cardiovascular event (MCE) into low (0 or 1 point), intermediate (2 or 3 points) or high (4, 5 or 6 points).

Investigator's hypothesis is that the HAR score could be entrusted to MRA, to enable them to optimize the prioritization of patients calling with non-traumatic chest pain, by qualifying low-risk chest pain calls on the one hand, which could be prioritized in P2 SNP, and high-risk calls on the other, making it possible to anticipate the dispatch of an emergency service.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (≥ 18 years)
* Calling Center 15 from 49, 72 or 37
* Expressing non-traumatic chest pain, even if this is not the main reason for seeking help.

Exclusion Criteria:

* Treatment in departments other than 49, 72 and 37
* Taken in charge in an emergency department of a private facility in the 49, 72 and 37 départements
* Poor understanding of the French language
* Non-affiliated or non-beneficiary of a social security scheme
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person subject to a legal protection measure
* Person unable to express his/her non-opposition.
* Follow-up at Day 30 impossible for any reason
* Person having expressed his/her opposition to the collection of his/her data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients calling center 15 for chest pain
Sampling Method: Non-Probability Sample
Enrollment: 796 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of major cardiovascular events | 30 days
  Number of major cardiovascular events is measured by presence of Death from cardiological causes, Type 1 or 2 myocardial infarction, Percutaneous coronary intervention, Surgical coronary bypass surgery

SECONDARY OUTCOMES:
Performance of the HAR Score: Sensitivity, Specificity, and Comparison Between EMR and MRA | From Day 0 to Day 30
  Sensitivity, specificity, likelihood ratios of the HAR score at different decision thresholds and the area under the ROC curve, as well as reclassification rates between the evaluation of the HAR score by the EMR (Emergency Medical Dispatcher) and the MRA (Medical Regulation Assistant)
Comparaison between rescue resources decided and predicted by the HAR score | From Day 0 to Day 30
  The proportion of rescue resources (SMUR - VSAV...) that would have been decided according to the HAR score (≥ 4 points) compared to the proportion of rescue resources actually decided upon
Time delta between the end of the MRA's score suggesting the dispatch of equipment (HAR score ≥ 4 points) and the actual decision to dispatch equipment in the current situation. | From Day 0 to Day 30
Area under the ROC curve and Delong-Delong test | From Day 0 to Day 30

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Le Mans, Le Mans
  - CHRU de Tours, Tours